CLINICAL TRIAL: NCT03188419
Title: Retrospective Study of the Breadth of Donor Options for Patients With Inherited Diseases Requiring Allogeneic Hematopoietic Stem Cell Transplant in the Era of Alternative Donor Transplants Using Post-Transplantation Cyclophosphamide
Brief Title: Breadth of Donor Options for People With Inherited Diseases Requiring Allogeneic Hematopoietic Stem Cell Transplant in the Era of Alternative Donor Transplants Using Post-Transplantation Cyclophosphamide
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917104; 17-C-N104
Record Dates: First submitted 2017-06-14; First posted 2017-06-15 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Primary T-cell Immunodeficiency Disorders; Common Variable Immunodeficiency
Keywords: Prospective Donors; Immunodeficiency
MeSH Terms: conditions — T cell immunodeficiency primary; Common Variable Immunodeficiency; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Retrospective chart review of patients with inherited immunodeficiency diseases requiring allogeneic hematopoietic stem cell transplant (allo HSCT)

SUMMARY:
Background:

People who have certain immune system diseases often need a procedure called allo HSCT. This is short for allogeneic hematopoietic stem cell transplant. This might cure people with these diseases. Many people who need allo HSCT need donors who are relatives with similar genes. But the disease may also affect those in the donor pool. This may mean there are fewer options for people with inherited diseases. Researchers want to collect data on how transplant candidates and their donors are found.

Objective:

To find out how genetic diseases and the ways they are inherited affect the breadth of options for allo HSCT donors.

Eligibility:

Records from studies that have already been done. These will be for people ages 4 and older who were evaluated for allo HSCT or to be donors.

Design:

Participants already signed a consent form for their records to be shared.

Researchers will study the participant data.

Data will be stored in an electronic system. Researchers will use passwords to protect the data.

DETAILED DESCRIPTION:
This protocol is a retrospective review of donor search results for patients with inherited immunodeficiency diseases requiring allogeneic hematopoietic stem cell transplant (allo HSCT).

The study will involve collecting information related to the donor search for transplant candidates and their prospective donors, using records in CRIS, Crimson, the HLA lab, and records in the transplant coordinator office (such as shipping logs of HLA typing kits). The study will not involve the use of specimens or participant contact.

The participants whose records will be reviewed will be those who were evaluated for allo HSCT or donation on an NIH primary immunodeficiency transplant protocol at a time when haplo donors were eligible (March 30, 2012 to present for GATA2, January 1, 2015 for CGD, October 6, 2015 to present for 16-C-0003, and May 21, 2014 to present for DOCK8).

The Principal Investigators on the included protocols have granted permission to conduct this study and have verified that none of the original protocols or informed consent documents preclude such a review of clinical data.

ELIGIBILITY:
* Data Analysis Only

Ages: 4 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective chart review of patients who with inherited immunodeficiency diseases requiring allogeneic hematopoietic stem cell transplant (allo HSCT)at the NIH Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
To determine the impact of genetic diseases and their modes of inheritance on the breadth of allo HSCT donor options | 1 year
  To determine the impact of genetic diseases and their modes of inheritance on the breadth of allo HSCT donor options

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hsieh MM, Kang EM, Fitzhugh CD, Link MB, Bolan CD, Kurlander R, Childs RW, Rodgers GP, Powell JD, Tisdale JF. Allogeneic hematopoietic stem-cell transplantation for sickle cell disease. N Engl J Med. 2009 Dec 10;361(24):2309-17. doi: 10.1056/NEJMoa0904971. PMID 20007560
- [Background] Gragert L, Eapen M, Williams E, Freeman J, Spellman S, Baitty R, Hartzman R, Rizzo JD, Horowitz M, Confer D, Maiers M. HLA match likelihoods for hematopoietic stem-cell grafts in the U.S. registry. N Engl J Med. 2014 Jul 24;371(4):339-48. doi: 10.1056/NEJMsa1311707. PMID 25054717